CLINICAL TRIAL: NCT05625321
Title: Community-Based Strategies to Reduce Cardiometabolic Disease in the Deep South
Brief Title: Stepping Into Lifestyle Changes
Acronym: SILC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Mississippi Medical Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Monica L Baskin, Adjunct Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 300009477; P50MD017338 (NIH)
Record Dates: First submitted 2022-11-02; First posted 2022-11-22 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Overweight and Obesity; Pre-Diabetes; High Blood Pressure
MeSH Terms: conditions — Overweight; Obesity; Glucose Intolerance; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational Group Weight Loss Classes (Active Comparator): Participants will participate in a 12-month weight loss program, taught by lay health educators, and designed to promote and encourage healthy weight loss, dietary changes, and increased physical activity. Participants will attend 90-minute sessions weekly for 6 months, bi-weekly for 3 months, and monthly for 3 months.
  Interventions: Behavioral: Educational Group Weight Loss Classes
- Educational Group Weight Loss Classes PLUS Home Gardening Intervention (Experimental): Participants will receive the educational group weight loss classes PLUS a home gardening intervention. The gardening intervention will be led by local Master Gardeners (MGs) who will help guide participants in setting-up and maintaining their garden.
  Interventions: Behavioral: Educational Group Weight Loss Classes; Behavioral: Home Gardening Intervention

INTERVENTIONS:
Behavioral: Educational Group Weight Loss Classes — Participants will be provided with educational materials on weight loss, and have opportunities to increase their exercise and make changes to their diet.
Behavioral: Home Gardening Intervention — Participants will receive tools to establish their own home garden, increasing their access to fresh fruits and vegetables.
  Arms: Educational Group Weight Loss Classes PLUS Home Gardening Intervention

SUMMARY:
The purpose of this study is to promote healthy weight loss among African American women, age 30 or older, who are pre-diabetic and/or have high blood pressure and who live, work, or worship in select rural communities throughout Alabama and Mississippi. The goal of the study is to help reduce the burden of obesity, diabetes, and high blood pressure for these women and to collect information on the reach, effectiveness, adoption, implementation, maintenance, and cost effectiveness of our two evidence-base weight loss programs.

DETAILED DESCRIPTION:
This study leverages two evidence-based interventions (EBIs) that have been culturally-adapted for the target population and have previously achieved clinically-relevant weight loss and other clinical outcomes (educational group weight loss intervention) along with improvements in diet and physical activity (home gardening intervention). Combining these EBIs addresses multiple domains (behavioral, personal environment, sociocultural) and levels (individual, interpersonal, community) of influence on risk factors for obesity and other cardiometabolic diseases prevalent in the Deep South. These interventions, delivered by local lay staff and non-academic partners, have a high potential for sustainability; however, there is a need to further evaluate the external validity and implementation-related barriers and facilitators to maximize reach, adoption and implementation. The investigators will employ a pragmatic, multilevel, cluster-randomized, type 1 hybrid effectiveness-implementation trial. A total of 264 Black women (age ≥ 30 years) with overweight or obesity and pre-diabetic or hypertensive from 12 rural counties (6 Alabama, 6 Mississippi) will receive either the combined educational group weight loss intervention plus a home gardening intervention or the educational group weight loss classes alone. The specific aims are to compare interventions on: (1) primary outcomes related to implementation effectiveness (reach, adoption, maintenance of health behaviors), (2) secondary outcomes on clinical effectiveness, and (3) cost effectiveness. Findings will inform discussions with coalition partners to achieve our long-term goal of widely disseminating and sustaining multi-level interventions to reduce the multiple chronic disease burden and health disparities in the Deep South.

ELIGIBILITY:
Inclusion Criteria:

* self-identifies as Black and/or African American
* ≥ 30 years old
* a measured BMI >25 kg/m2 and at least one other cardiometabolic risk factor (physician diagnosis of pre-diabetes and/or hypertension within past 2 years)
* lives, works, or worships in one of the 12 intervention communities and expresses no intentions to move outside of that community in the 18 months following enrollment
* a willingness to participate in the study for the 18-months duration.

Exclusion Criteria:

* being or planning to become pregnant during the 18-month study duration
* a baseline blood pressure and/or glucose that is outside of the normal range and a medical provider does not provide clearance to participate
* medical contraindications

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight | 0, 6, and 12 months
  Changes in Weight, measured in pounds
BMI | 0, 6, and 12 months
  Changes in BMI, calculated as a person's weight in kilograms divided by the square of height in meters
Waist Circumference | 0, 6, and 12 months
  Changes in waist circumference, measured in centimeters
Dietary Intake | 0, 6, and 12 months
  Changes in diet, measured using a questionnaire

SECONDARY OUTCOMES:
Diastolic and Systolic Blood Pressure | 0, 6, and 12 months
  Changes in values over time, using a calibrated automatic sphygmomanometer and following NHLBI protocols
Fasting Glucose | 0, 6, and 12 months
  Changes in glucose readings, collected by finger-stick
Cholesterol Levels | 0, 6, and 12 months
  Changes in LDL and HDL values/ratio, collected by finger-stick
Physical Activity | 0, 6, and 12 months
  Changes in physical activity, measured by the International Physical Activity Questionnaire (IPAQ).
  For the IPAQ survey, participants will be asked to indicate if they have completed low (sitting or walking) levels of activity, moderate levels of activity, and/or high levels of activity in the last 7 days.They will also be asked to provide the number of days they do each activity and the time, in minutes, they spend doing the activity.
Physical Activity | 0, 6, and 12 months
  Changes in physical activity, measured by the Stanford Leisure Time Activity Categorical Item (L-cat).
  The L-Cat is categorical and responses range from 1-6 with 1 indicating little to no physical activity, and 6 indicating vigorous activity for 5 or more days a week.
Perceived Quality of Life | 0, 6, and 12 months
  Changes in Quality of Life as measured by the EuroQol-5 Dimension survey (EQ-5D-5L). Condition states range from 1-5 with 1 meaning the participant has no problems or symptoms and 5 meaning they have are unable to perform the activity or are extremely impacted by the condition. Self reported health is measured on a 1 to 100 scale with 1 being the worst possible health and 100 being the best possible health.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Baskin, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No